CLINICAL TRIAL: NCT01448252
Title: Autologous T Cell Vaccination With Line Specific for 9 Myelin Peptides in Patients With Progressive / Relapsing Multiple Sclerosis
Brief Title: T Cell Vaccination in Patients With Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Dimitrios Karussis, Head, Multiple Sclerosis Center, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCV-HMO-CTIL; 27-15.15.00 (Other: Hmo)
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Multiple Sclerosis
Keywords: T cell vaccination; Immunotherapy; Tolerance; safety; clinical efficacy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TCV (Active Comparator): multiple T cell vaccinations against nine myelin peptides at days 1, 30, 90, 180
  Interventions: Biological: T cell vaccination
- Placebo (Sham Comparator): saline injections subcutaneously at the same 4 time points with active treatment
  Interventions: Biological: multiple (4 autologous subcutaneous T cell vaccinations with T cell lines reactive to nine myelin peptides)

INTERVENTIONS:
Biological: multiple (4 autologous subcutaneous T cell vaccinations with T cell lines reactive to nine myelin peptides) — multiple (4 autologous subcutaneous T cell vaccinations with T cell lines reactive to nine myelin peptides at days 1, 30,90,180
  Other Names: multiple subcutenous injections of saline at days 1, 30,90,180.
  Arms: Placebo
Biological: T cell vaccination — Multiple injections of autologous T cell lines reactive to 9 myelin peptides.
  Arms: TCV

SUMMARY:
This is a double blind phase I-II clinical trial with multiple autologous T cell vaccinations using T cell lines reactive to 9 different myelin peptides of MBP, MOG and PLP, in patients with relapsing progressive Multiple Sclerosis.

DETAILED DESCRIPTION:
This trial is a phase I/II double-blind controlled clinical trial designed to evaluate the safety and clinical efficacy of multiple autologous T-cell vaccinations (on days 1, 30, 90 and 180) in progressive MS patients which showed severe progression/deterioration in the functional status (at least, one degree in the EDSS scale) during the last year, or at least one severe relapse. The patients will be from our MS clinic and will be randomized (by computer) into two groups according to: age, disease duration, disease severity and progression rate. One group (2/3 of the patients) will receive the active treatment, i.e. TCV, and the other group (1/3 of the patients) will receive sham treatment (injection of sterile normal saline). The treating nurse, the treating physician, the examining neurologist (the one who will perform the neurological evaluation) and the patient will be blinded for the treatment.

OBJECTIVES AND SIGNIFICANCE OF THE TRIAL

A. To develop a new cell therapeutic modality for treating MS patients using attenuated autologous anti-MBP, anti-PLP and anti-MOG autoreactive T-cells as vaccines. The immune response induced by this vaccination will be directed specifically against the T-cells attacking the patient's nerve system (specifically the myelin sheath).

B. To study and characterize these autoreactive T-cells in MS patients. The number and function of such cells in the course of the relapse of the disease, as well as during the periods of remissions, will be studied.

C. To study the clinical efficacy of T-cell vaccination with attenuated anti-MBP and anti-MOG autologous T-cells on MS. The parameters to be examined will include: change in the disability status (by the EDSS disability scale, as well as by ambulation index and several other functional tests), the change in the relapse rate and in the timed 10-meters walking test, the PASAT test and the 9-hole peg test. MRI parameters will represent additional endpoints and will include: the changes in the total burden of the disease and in the quantity of irreversible damage (cortical atrophy and axonal loss). In addition, the effects of this treatment on the immune responses (i.e. number and proportion of activated lymphocytes, number and proportion of anti-myelin reactive lymphocytes in the peripheral blood and IgG antibody levels in the cerebrospinal fluid) will be evaluated in the treated MS patients.

The significance and importance of the study are outlined as follows:

1. It offers a new approach for the treatment of MS.
2. This approach has the advantage of being devoid of toxic or general immunosuppressive effects.
3. The study will pave the way for further studies that will improve our understanding of the mechanisms of the host immune response in MS and of the involvement of the MBP, PLP and MOG myelin proteins in the initiation of the auto-reactive immune response and of clinical MS.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite MS (according to Poser's criteria) of the relapsing-progressive type (RPMS).
2. Age: 18-60.
3. EDSS: 3.0 to 7.0.
4. Disease duration: > 1 year.
5. Evidence of disease progression of 1 degree in the EDSS scale, or at least two severe relapses (requiring hospitalization and treatment) during the year prior to inclusion.
6. MRI of the brain with at least 5 lesions in the white matter (T2 imaging).
7. Failure to benefit from other existing treatments according to the guidelines of the Israeli Ministry of Health.

Exclusion Criteria:

1. Patients with other systemic active disease.
2. Patients who had been treated with immunosuppressive drugs during the 3-6 months depending on the cytotoxicity of the medication used prior to the inclusion.
3. Patients who previously received cellular immunotherapy or who are participating in other experimental protocols.
4. Pregnancy; Pregnant women or women who do not use efficacious contraception (oral contraception, or intra-uterine device).
5. Patients with an additional autoimmune condition unrelated to MS or significant allergy.
6. Patients who cannot fully understand the treatment protocol or are unable to sign the informed consent, or in whom the clinician believes that a follow-up period of at least 12 months will not be possible.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-05; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
EDSS changes | one year
  Follow up in changes in the EDSS score
Relapse rate of MS | one year follow up
  recording of the relapses of MS during the year of the study and the prior to the study
PASAT test | one year
  recording of the performance in the PASAT test during the one year of the study
Nine hole PEG test | one year
  recording of the performance in the Nine hole PEG test test during the one year of the study
timed ten meter walking | one year
  recording of the performance in the timed ten meter walking test during the one year of the study

SECONDARY OUTCOMES:
Quantitative MRI evaluation | one year
  the burden of T2 lesions load, of the hypo-intense T1 lesions, of the Gadolinium enhancing lesions and of the brain atrophy will be evaluated at the end of the study and compared to the baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karussis, Prof., Principal Investigator — Hadassah Medical Organizatin; Rivka Abulafia-Lapid, PhD, Study Director — Hadassah Medical Organization
Locations (1):
- Dept of Neurology,Hadassah ein-Kerem, Jerusalem, Israel

REFERENCES:
- [Derived] Karussis D, Shor H, Yachnin J, Lanxner N, Amiel M, Baruch K, Keren-Zur Y, Haviv O, Filippi M, Petrou P, Hajag S, Vourka-Karussis U, Vaknin-Dembinsky A, Khoury S, Abramsky O, Atlan H, Cohen IR, Abulafia-Lapid R. T cell vaccination benefits relapsing progressive multiple sclerosis patients: a randomized, double-blind clinical trial. PLoS One. 2012;7(12):e50478. doi: 10.1371/journal.pone.0050478. Epub 2012 Dec 14. PMID 23272061